CLINICAL TRIAL: NCT02734069
Title: Impact of Fat-free Mass in the Carboplatin Calculated Dose and Chemotherapeutic Toxicity in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Impact of Fat-free Mass in the Carboplatin Calculated Dose and Chemotherapeutic Toxicity in Patients With Advanced NSCLC
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of the Thoracic Oncology Unit and Laboratory of Experimental Oncology, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: INCAN/TOX/CBP
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Sarcopenia; Toxicity
Keywords: carboplatin
MeSH Terms: conditions — Lung Neoplasms; Sarcopenia | interventions — Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sarcopenic: Patients with sarcopenia (evaluated according to CT scans) will be followed up through treatment with carboplatin for identification of any toxicity grade 3 or 4 (Common Terminology Criteria of Adverse Events)
  Interventions: Drug: Carboplatin
- Non Sarcopenic: Patients without sarcopenia (evaluated according to CT scans) will be followed up through treatment with carboplatin for identification of any toxicity grade 3 or 4 (Common Terminology Criteria of Adverse Events)
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Patients will receive carboplatin according to the carboplatin area under the curve dose calculation for 2 cycles to evaluate toxicity.
  Other Names: CARBOPLAT

SUMMARY:
This study evaluate the association of body composition (mainly free-fat mass), clinical and biochemical parameters with development of toxicity in patients under treatment with Carboplatin/Paclitaxel in advanced NSCLC.

DETAILED DESCRIPTION:
BACKGROUND

Lung cancer (LC) is the leading cause of cancer deaths worldwide, are attributed about 13% of all new cases of cancer and accounts for 19.4% of deaths from malignancies. In Mexico, this cancer is also the leading cause of death in malignant neoplasias. One of the reasons attributable the high mortality from this disease is that most cases are detected in advanced stages and this depends prognosis and treatment. Within the classification of LC the most prevalent is the Non Small Cell Lung Cancer (NSCLC); for which the considered first-line standard treatment is palliative cytotoxic chemotherapy, as the combination of carboplatin with paclitaxel and in the other hand one of the most recent combinations Carboplatin with Pemetrexed.

Malnutrition may affect 80% of patients with advanced cancer and is associated with up to 20% of deaths, with an increased risk in the development of complications and mortality and can extend the hospital stay up to 90%, increasing the cost of treatment in a 35-75%. Similarly, in a previous study at INCan, the degree of malnutrition in patients with LC was associated with cytotoxic chemotherapy toxicity and poorer prognosis and poorer quality of life. Sarcopenia is also a phenomenon commonly observed in patients with LC, there has been a prevalence of 61% and 31% in men and women respectively.

Carboplatin dose that is administered to the patient is calculated by the Calvert formula, this requires the calculation of glomerular filtration rate (GFR). There are various quantified and estimated methods to calculate GFR; however the validated and most commonly used is estimated by the Cockroft-Gault formulae. It is known that due to various factors, variables required for calculation (as creatinine) could be modify the result, may became unreliable, it is why it is important to consider changes in body composition of NSCLC patients with sarcopenia.

HYPOTHESIS:

Sarcopenia participants receive a 20% more dose of Carboplatin per Free Fat Mass (kg / mg) than those without sarcopenia.

Sarcopenic patients, have more severe toxicity related to chemotherapy than those without sarcopenia.

METHODOLOGY:

NSCLC patients with advanced NSCLC (inoperable stage III or IV ) will be included.

Clinicopathological baseline of patients such as age, sex, stage, ECOG, weight, height, body composition, Subjective Global Assessment, frequency of food consumption, albumin, hemoglobin, hematocrit, glomerular filtration rate, carboplatin administered dosage, quality of life, etc.

A subsequent follow-up evaluation will be made after 1st and 2nd cycle of treatment to assess toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSCLC Stage IV (stratification according to the American Joint Committee on Cancers - 7th edition)
* Candidates for treatment with carboplatin plus paclitaxel 1st line
* Performance status (ECOG 0-2)
* Laboratory studies that demonstrate adequate renal, hepatic and hematologic function (blood chemistry and blood count)
* Normal renal ultrasound prior to initiation of treatment

Exclusion Criteria:

* Patients with renal impairment (KDOQI 3-5)
* Patients who do not have computed tomography study at baseline
* Uncontrolled blood pressure (> 140 mmHg)
* Uncontrolled diabetes (> 130 mg / dL)
* Obstruction in kidney (s) or ureter (s)
* Dehydrated patients
* Patients with high consumption of NSAIDs (aspirin, ibuprofen, etc.> 1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC, as candidates for the first line chemotherapy regimen of carboplatin / paclitaxel or Carboplatin / Pemetrexed
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Three weeks after the application of chemotherapy to detect changes from Baseline
  Determine if the dose of carboplatin-based chemotherapy in patients according to the amount of fat-free mass is directly associated with toxicity
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Six weeks after the application of chemotherapy to detect changes from Baseline
  Determine if the dose of carboplatin-based chemotherapy in patients according to the amount of fat-free mass is directly associated with toxicity

SECONDARY OUTCOMES:
Compare different formulas to calculate Glomerular Filtration Rate taking as gold standard cystatin c | Basal evaluation
  Calculate the glomerular filtration rate given the amount of fat-free mass (MSA-eCrCl) and correlate with cystatin C and formulas as Cockroft-Gault, Levey, The Modification of Diet in Renal Disease (MDRD) and Chronic kidney disease epidemiology collaboration (CKD-EPI).

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, MSc, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Ruiz-Godoy L, Rizo Rios P, Sanchez Cervantes F, Osornio-Vargas A, Garcia-Cuellar C, Meneses Garcia A. Mortality due to lung cancer in Mexico. Lung Cancer. 2007 Nov;58(2):184-90. doi: 10.1016/j.lungcan.2007.06.007. Epub 2007 Jul 30. PMID 17659812
- [Background] Cullen MH, Billingham LJ, Woodroffe CM, Chetiyawardana AD, Gower NH, Joshi R, Ferry DR, Rudd RM, Spiro SG, Cook JE, Trask C, Bessell E, Connolly CK, Tobias J, Souhami RL. Mitomycin, ifosfamide, and cisplatin in unresectable non-small-cell lung cancer: effects on survival and quality of life. J Clin Oncol. 1999 Oct;17(10):3188-94. doi: 10.1200/JCO.1999.17.10.3188. PMID 10506617
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Gronberg BH, Bremnes RM, Flotten O, Amundsen T, Brunsvig PF, Hjelde HH, Kaasa S, von Plessen C, Stornes F, Tollali T, Wammer F, Aasebo U, Sundstrom S. Phase III study by the Norwegian lung cancer study group: pemetrexed plus carboplatin compared with gemcitabine plus carboplatin as first-line chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2009 Jul 1;27(19):3217-24. doi: 10.1200/JCO.2008.20.9114. Epub 2009 May 11. PMID 19433683
- [Background] Gordon JN, Green SR, Goggin PM. Cancer cachexia. QJM. 2005 Nov;98(11):779-88. doi: 10.1093/qjmed/hci127. Epub 2005 Oct 7. PMID 16214835
- [Background] Ottery FD. Cancer cachexia: prevention, early diagnosis, and management. Cancer Pract. 1994 Mar-Apr;2(2):123-31. PMID 8055014
- [Background] Muscaritoli M, Bossola M, Aversa Z, Bellantone R, Rossi Fanelli F. Prevention and treatment of cancer cachexia: new insights into an old problem. Eur J Cancer. 2006 Jan;42(1):31-41. doi: 10.1016/j.ejca.2005.07.026. Epub 2005 Nov 28. PMID 16314085
- [Background] Sanchez-Lara K, Turcott JG, Juarez E, Guevara P, Nunez-Valencia C, Onate-Ocana LF, Flores D, Arrieta O. Association of nutrition parameters including bioelectrical impedance and systemic inflammatory response with quality of life and prognosis in patients with advanced non-small-cell lung cancer: a prospective study. Nutr Cancer. 2012;64(4):526-34. doi: 10.1080/01635581.2012.668744. Epub 2012 Apr 10. PMID 22489794
- [Background] Baracos VE, Reiman T, Mourtzakis M, Gioulbasanis I, Antoun S. Body composition in patients with non-small cell lung cancer: a contemporary view of cancer cachexia with the use of computed tomography image analysis. Am J Clin Nutr. 2010 Apr;91(4):1133S-1137S. doi: 10.3945/ajcn.2010.28608C. Epub 2010 Feb 17. PMID 20164322
- [Background] Calvert AH, Newell DR, Gumbrell LA, O'Reilly S, Burnell M, Boxall FE, Siddik ZH, Judson IR, Gore ME, Wiltshaw E. Carboplatin dosage: prospective evaluation of a simple formula based on renal function. J Clin Oncol. 1989 Nov;7(11):1748-56. doi: 10.1200/JCO.1989.7.11.1748. PMID 2681557
- [Background] Nannan Panday VR, van Warmerdam LJ, Huizing MT, Ten Bokkel Huinink WW, Vermorken JB, Giaccone G, Veenhof CH, Schellens JH, Beijnen JH. Carboplatin dosage formulae can generate inaccurate predictions of Carboplatin exposure in carboplatin/paclitaxel combination regimens. Clin Drug Investig. 1998;15(4):327-35. doi: 10.2165/00044011-199815040-00009. PMID 18370488
- [Background] Hudson JQ, Owens HM, Fleckenstein JF, Loveless VS, Krauss AG, Hak LJ. Performance of methods to assess kidney function in a predominantly overweight sample of patients with liver disease. Ren Fail. 2013;35(2):249-56. doi: 10.3109/0886022X.2012.745786. Epub 2012 Nov 26. PMID 23176438
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Botev R, Mallie JP, Wetzels JF, Couchoud C, Schuck O. The clinician and estimation of glomerular filtration rate by creatinine-based formulas: current limitations and quo vadis. Clin J Am Soc Nephrol. 2011 Apr;6(4):937-50. doi: 10.2215/CJN.09241010. Epub 2011 Mar 31. PMID 21454722
- [Background] Ekhart C, Rodenhuis S, Schellens JH, Beijnen JH, Huitema AD. Carboplatin dosing in overweight and obese patients with normal renal function, does weight matter? Cancer Chemother Pharmacol. 2009 Jun;64(1):115-22. doi: 10.1007/s00280-008-0856-x. Epub 2008 Nov 7. PMID 18989671
- [Background] Kaag D. Carboplatin dose calculation in lung cancer patients with low serum creatinine concentrations using CKD-EPI and Cockcroft-Gault with different weight descriptors. Lung Cancer. 2013 Jan;79(1):54-8. doi: 10.1016/j.lungcan.2012.10.009. Epub 2012 Nov 4. PMID 23131495